CLINICAL TRIAL: NCT00827723
Title: Makuuchi Versus Barcelona Clinic of Liver Cancer Criteria in Cirrhotic Patients With Hepatocellular Carcinoma. Does Etiology of Cirrhosis Influence the Relationship Between the Portal Pressure and Quantitative Tests of Liver Function?
Brief Title: Indocyanine Green and Portal Pressure in Viral and Alcoholic Cirrhotic Patients With Hepatocarcinoma
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Nicolas DEMARTINES, professor of surgery, University of Lausanne Hospitals
Other Study IDs: 251/08
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Carcinoma, Hepatocellular; Alcoholic Cirrhosis; Viral Cirrhosis; Postoperative Hepatic Failure
Keywords: Hepatic functional reserve; Hepatocellular carcinoma (HCC); Indocyanine Green retention rate at 15 minutes (ICG-R15'); Portal Pressure (PP); Hepatic Portal Venous Gradient (HPVG); Alcoholic and Viral Cirrhosis; Makuuchi criteria; Barcelona Clinic of Liver Cancer (BCLC); Hepatic resection
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis, Alcoholic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Alcoholic: Alcoholic cirrhotic patient with resectable hepatocellular carcinoma
- Viral: Viral cirrhotic patient with resectable hepatocellular carcinoma

SUMMARY:
The aim of the investigators' study is to elucidate the relationship between a functional liver test (e.g., ICG) and the PREOPERATIVE value of portal hypertension in the patients with impaired liver function from alcoholic and non-alcoholic aetiologies. Alcoholic and viral cirrhosis present important differences in terms of cellular mechanisms responsible for the disease progression with a distinct and unique gene expression pattern that regulates the type of inflammatory response. These differences probably influence the hepatic functional reserve and the onset of portal hypertension at a comparable clinical and biological level of derangement and the investigators may expect significant differences in the recovery from hepatectomy.

The investigators' hypothesis is that at a comparable ICGR-15 rate non-viral cirrhotic liver presents higher portal pressure values and the investigators also argue that alcoholic cirrhotic patients would tolerate a larger hepatic resection than would viral cirrhotic do.

ELIGIBILITY:
Inclusion Criteria:

* resectable or amenable to resection HCC in cirrhotic child A patients of alcoholic or viral etiology

Exclusion Criteria:

* cirrhosis Child-Pugh B
* absence of patient consent
* psychiatric pathology

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
concordance rate between ICGR-15 and Portal Pressure values in patients with resectable HCC and cirrhosis Child A from alcoholic and non-alcoholic origin. | 1 year

SECONDARY OUTCOMES:
postoperative liver failure. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Diana Michele, MD, Principal Investigator — CHUV University Hospital of Lausanne; Halkic Nermin, PD, Study Director — CHUV University Hospital of Lausanne; Demartines Nicolas, Professeur, Study Chair — CHUV University Hospitals of Lausanne
Locations (1):
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Yamazaki S, Takayama T. Surgical treatment of hepatocellular carcinoma: evidence-based outcomes. World J Gastroenterol. 2008 Feb 7;14(5):685-92. doi: 10.3748/wjg.14.685. PMID 18205256
- [Background] Imamura H, Seyama Y, Kokudo N, Maema A, Sugawara Y, Sano K, Takayama T, Makuuchi M. One thousand fifty-six hepatectomies without mortality in 8 years. Arch Surg. 2003 Nov;138(11):1198-206; discussion 1206. doi: 10.1001/archsurg.138.11.1198. PMID 14609867
- [Background] Torzilli G, Makuuchi M, Inoue K, Takayama T, Sakamoto Y, Sugawara Y, Kubota K, Zucchi A. No-mortality liver resection for hepatocellular carcinoma in cirrhotic and noncirrhotic patients: is there a way? A prospective analysis of our approach. Arch Surg. 1999 Sep;134(9):984-92. doi: 10.1001/archsurg.134.9.984. PMID 10487594
- [Background] Llovet JM, Burroughs A, Bruix J. Hepatocellular carcinoma. Lancet. 2003 Dec 6;362(9399):1907-17. doi: 10.1016/S0140-6736(03)14964-1. PMID 14667750
- [Background] Bruix J, Castells A, Bosch J, Feu F, Fuster J, Garcia-Pagan JC, Visa J, Bru C, Rodes J. Surgical resection of hepatocellular carcinoma in cirrhotic patients: prognostic value of preoperative portal pressure. Gastroenterology. 1996 Oct;111(4):1018-22. doi: 10.1016/s0016-5085(96)70070-7. PMID 8831597
- [Derived] Kobayashi K, Uldry E, Kokudo T, Cristaudi A, Kawaguchi Y, Shirata C, Yamaguchi T, Dormond O, Duran R, Hasegawa K, Demartines N, Halkic N. Correlation Between Portal Pressure and Indocyanine Green Retention Rate is Unaffected by the Cause of Cirrhosis: A Prospective Study. World J Surg. 2021 Aug;45(8):2546-2555. doi: 10.1007/s00268-021-06111-6. Epub 2021 Apr 23. PMID 33891139